CLINICAL TRIAL: NCT05827965
Title: Ramadan Fasting in Secondary Adrenal Insufficiency Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Rabta (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, Professor, Hopital La Rabta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1/2023
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Secondary Adrenal Insufficiency; Fasting, Intermittent
Keywords: secondary adrenal insufficiency; intermittent fasting; complications; education; glucocorticoid replacement therapy; lifestyle
MeSH Terms: conditions — Intermittent Fasting | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: before and after education and drug adjustement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with secondary adrenal insufficiency (Experimental): education and treatment adjustment
  Interventions: Behavioral: education and drug adjustement

INTERVENTIONS:
Behavioral: education and drug adjustement — education of the patients (lifestyle) and adjustement of glucocorticoid replacement schedule

SUMMARY:
Intermittent Ramadan fasting was associated with a risk of complications in patients with adrenal insufficiency. A risk stratification with recommendations (lifestyle and drug adjustment) for fasting in these patients has been recently published. So, this prospective interventional study was carried out to evaluated these recommendations. Patients with secondary adrenal insufficiency and willing to fast Ramadan were included. Before Ramadan, patients underwent a clinical examination and were educated for lifestyle measures and the schedule of glucocorticoid replacement therapy was adjusted. The occurrence of complications and the number of fasted days during the month of Ramadan 2023 were reported and compared with those of Ramadan 2022.

DETAILED DESCRIPTION:
Intermittent fasting during the month of Ramadan is one of the five pillars of Islam and a sacred ritual for Muslims. Patients with chronic diseases seek advice from their physician and insist on fasting. A former study showed that 76.7% of adrenal insufficiency patients were exempted from fasting and 50.5% of them fasted against the advice of their physician. Few studies have assessed the risk of complications in adrenal insufficiency patients. The most frequently reported complications were asthenia (88.5%), signs suggestive of dehydration (49.2%), intense thirst (32.8%), and signs of hypoglycaemia (18%). Hypoglycaemia was detected by 24 hour-continuous glucose monitoring in 10% of fasting patients with secondary adrenal insufficiency (SAI). These complications were more frequent in patients with insufficient knowledge of the disease. A literature review was published 2021 and a risk stratification of patients with adrenal insufficiency and recommendations for patient education and therapeutic adjustment were proposed. However, no study has evaluated the effect of these measures on Ramadan fasting in SAI.

The objectives were to:

1. compare the number of fasted days and the prevalence of complications during Ramadan fasting before (2022) and after therapeutic education and treatment adjustment (2023) in patients with SAI.
2. determine the factors associated with complications during Ramadan fasting in SAI.

Methods:

Before the month of Ramadan 2023, patients meeting the inclusion criteria were enrolled. All patients signed a written informed consent.

During the first visit, the following data were recorded:

* gender, age, medical and surgical history, current treatments, medication schedule, the 2022 fast (number of fasted days, complications (type, days, time, break of the fast for a complication)).
* weight, height, lying and standing blood pressure.
* Some data were taken from the medical file: other affected pituitary axes, etiology of the SAI, results of the insulin hypoglycaemia test if performed (baseline cortisol, peak level, peak time, area under the curve), plasma creatinine.

Subsequently, patient education (the particularities of the disease, the risks and lifestyle measures) and therapeutic adjustments were performed according to the recommendations published by Chihaoui et al in Endocrine, 2021.

Throughout the month of Ramadan 2023, patients filled in forms indicating for the fasted days: dinner time, shour time, sleep time, unusual physical activity, treatment schedule, occurrence of complications: type, time, break of the fast for a complication.

Throughout the study, regular telephone contact with one of the investigators was performed for any additional information, advice or therapeutic adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Secondary adrenal insufficiency patients
* Substituted with glucocorticoids for more than one year.
* Willing to fast during the month of Ramadan 2023

Exclusion Criteria:

* cardiac insufficiency,
* respiratory insufficiency,
* hepatic insufficiency,
* renal insufficiency (creatinine clearance < 60 ml/min/1.73m2),
* advanced neoplasia,
* undernutrition,
* diabetes insipidus,
* diabetes mellitus,
* neuro-psychiatric disease,
* infectious disease
* chronic inflammatory disease,
* hyperthyroidism,
* uncontrolled hypothyroidism,
* alcoholism,
* diuretic intake,
* glucocorticoid treatment for purposes other than substitution,
* treatment with enzyme inducers,
* pregnancy,
* breastfeeding
* consent withdrawn
* study discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
number of fasted days | one month
  change in the number of fasted days
prevalence of complications | one month
  change in the prevalece of complications

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital La Rabta, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the publication of this study

REFERENCES:
- [Background] Chihaoui M, Yazidi M, Oueslati I, Khessairi N, Chaker F. Intermittent fasting in adrenal insufficiency patients: a review and guidelines for practice. Endocrine. 2021 Oct;74(1):11-19. doi: 10.1007/s12020-021-02804-z. Epub 2021 Jul 2. PMID 34213700
- [Background] Chihaoui M, Chaker F, Yazidi M, Grira W, Ben Amor Z, Rejeb O, Slimane H. Ramadan fasting in patients with adrenal insufficiency. Endocrine. 2017 Jan;55(1):289-295. doi: 10.1007/s12020-016-1186-0. Epub 2016 Nov 23. PMID 27878773
- [Background] Chihaoui M, Grira W, Bettaieb J, Yazidi M, Chaker F, Rejeb O, Oueslati I, Feki M, Kaabachi N, Slimane H. The risk for hypoglycemia during Ramadan fasting in patients with adrenal insufficiency. Nutrition. 2018 Jan;45:99-103. doi: 10.1016/j.nut.2017.07.014. Epub 2017 Aug 3. PMID 29129244
- [Background] Hussain S, Hussain S, Mohammed R, Meeran K, Ghouri N. Fasting with adrenal insufficiency: Practical guidance for healthcare professionals managing patients on steroids during Ramadan. Clin Endocrinol (Oxf). 2020 Aug;93(2):87-96. doi: 10.1111/cen.14250. Epub 2020 Jun 15. PMID 32419166
- [Background] Chihaoui M, Mimita W, Oueslati I, Rejeb O, Ben Amor Z, Grira W, Yazidi M, Chaker F. Prednisolone or hydrocortisone replacement in patients with corticotrope deficiency fasting during Ramadan result in similar risks of complications and quality of life: a randomized double-blind controlled trial. Endocrine. 2020 Jan;67(1):155-160. doi: 10.1007/s12020-019-02082-w. Epub 2019 Sep 24. PMID 31552584
- [Derived] Mabrouk M, Chihaoui M, Sta J, Slimane CB, Oueslati I, Yazidi M, Chaker F. Ramadan Fasting Improves Health-Related Quality of Life in Patients With Secondary Adrenal Insufficiency: A Prospective Interventional Case-Control Study. Clin Endocrinol (Oxf). 2025 Oct;103(4):523-530. doi: 10.1111/cen.15286. Epub 2025 Jun 2. PMID 40452492
- [Derived] Chihaoui M, Mabrouk M, Oueslati I, Khessairi N, Chaker F, Yazidi M. Evaluation of therapeutic education on intermittent fasting in patients with secondary adrenal insufficiency: A clinical trial. Nutrition. 2025 Apr;132:112688. doi: 10.1016/j.nut.2025.112688. Epub 2025 Jan 14. PMID 39933257